CLINICAL TRIAL: NCT03954093
Title: Paired Transcranial Direct Current Stimulation/ Dorsal Root Ganglion Stimulation Trial
Brief Title: Paired Acute Invasive/Non-invasive Stimulation Trial
Acronym: PAINS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 13/SC/0298
Record Dates: First submitted 2019-05-10; First posted 2019-05-17 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2019-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sham stimulation (Sham Comparator)
  Interventions: Device: Transcranial direct current stimulation
- Motor cortex stimulation (Active Comparator)
  Interventions: Device: Transcranial direct current stimulation
- MEG-localized stimulation (Experimental)
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — tDCS produces hyper/hypopolarizing potentials in the cortex underlying the scalp electrodes and can increase/decrease the excitability of targeted brain regions.
  Other Names: tDCS

SUMMARY:
Chronic pain patients with implanted dorsal root ganglion stimulators will be randomized to receive transcranial direct current stimulation (tDCS) to the motor cortex, magneto-encephalographically (MEG) localized stimulation or sham stimulation to identify therapeutic efficacy of paired central and peripheral neuromodulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are willing and able to give consent to the study.
* Male or Female, aged 18 years or above with diagnoses of chronic pain.
* Treatment includes Spinal Cord Stimulation, Dorsal Root Ganglion stimulation, or peripheral analgesic stimulation.

Exclusion Criteria:

* Patients who do not wish to be in the study.
* Patients with metallic intracranial implants.
* Patients with extreme language barrier that cannot understand the purpose of the study despite the use of an interpreter

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Change in pain scores: 21-point pain scale rating | Immediately after 30 minutes of transcranial direct current stimulation
  21-point pain scale rating

SECONDARY OUTCOMES:
Changes in EEG recordings | Immediately after 30 minutes of transcranial direct current stimulation
  Changes in electrical fields of the cortex
Changes in Facial Expression Recognition Performance | Immediately after 30 minutes of transcranial direct current stimulation
  An emotional categorisation task to identify anti-depressant effects

CONTACTS AND LOCATIONS:
Overall Officials: Alex Green, FRCS, Principal Investigator — University of Oxford
Locations (1):
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Patient diagnoses and demographics will be shared but identities kept anonymous

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-28): https://cdn.clinicaltrials.gov/large-docs/93/NCT03954093/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-28): https://cdn.clinicaltrials.gov/large-docs/93/NCT03954093/ICF_001.pdf